CLINICAL TRIAL: NCT04796597
Title: Early Feasibility Study on Epios Leads
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wyss Center for Bio and Neuroengineering (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Device Feasibility
Other Study IDs: Epios
Record Dates: First submitted 2020-12-18; First posted 2021-03-15 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-arm (Experimental): Implantation of subcutaneous leads and connection to an external EEG amplifier
  Interventions: Device: Subcutaneous implantation of Epios sub-scalp leads

INTERVENTIONS:
Device: Subcutaneous implantation of Epios sub-scalp leads — The sub-scalp Epios Leads will be implanted by a trained neurosurgeon and will provide epicranial EEG recording of specific cortical areas identified by the neurologist.
  Other Names: Subcutaneous Epios leads insertion through tunneling toolkit with tear-away sheath

SUMMARY:
The Epios early feasibility study aims to explore the uses of novel sub-scalp lead devices in the detection of epileptic seizures. Epios leads are inserted subcutaneously through dedicated tunneling toolkits and have been designed for continuous EEG recording in inpatients.

This clinical investigation is part of a stepwise program to validate the entire Epios system and it starts with the validation of the Epios leads alone in this two steps study.

DETAILED DESCRIPTION:
According to the state of the art, epilepsy is defined as the spontaneous recurrence of seizures at random intervals. When epilepsy is drug refractory, management plans rely entirely on seizure self-reporting. However, it is now established that self-reports of seizure burdens are inaccurate. The reasons for this are multiple, but important ones include the fact that seizures can affect brain regions involved in awareness and memory, and that epilepsy patient can also have persistent cognitive deficits, so they do not recall having a seizure. EEG caps are the standard tool for monitoring brain waves, but this technology is typically used for less than an hour and rarely can be managed for a period of a week or so because of the need for continual technical interventions, like reapplying electrodes to the skin. Thus, there is no way to fill the gap in the ability to obtain monitoring of EEG for weeks, months or longer.

Given the unmet need for the objective monitoring of epileptic seizures in ambulatory patients, innovative solutions are under development.

The Epios device under investigation in this study consists in novel sub-scalp leads implanted between the scalp and the skull through an insertion tunneling toolkit for EEG monitoring in short-term conditions.

This clinical investigation is part of a stepwise program to validate the entire Epios system and it starts with the validation of the Epios leads alone in step 1 and step 2.

Step 1 is an intra-operative step only, where a 10-minute long EEG recording is performed using the Epios leads, after the patient has undergone general anesthesia for his/her clinically-indicated brain surgery. The study material is removed before skin closure and end of anesthesia.

Step 2 is an inpatient, short-term step, where, following clinically-indicated surgery for brain electrode implantation, the participants will stay in a continuous care unit. Clinical care and study recordings (with Epios subscalp leads) will be carried out in parallel. The Epios leads will remain implanted for the same length of time as the clinical electrodes: clinical EEG workups in epilepsy last one week at the clinical trial hospital, rarely two weeks, virtually never longer. In adherence to this approach, the implantation period of the investigational electrode in step 2 will be less than twenty one days (< 21 days).

Steps 1 and 2 will take 12 to 18 months in total. First participant-In is planned in January 2021 for step 1 and last participant-In is planned in July 2022.

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 18 years
* Informed Consent as documented by signature
* Neurosurgical patient, i.e. patient under surgical care who will undergo one of the following specific procedures:
* Step 1: Patient in the operating room undergoing clinically indicated brain surgery either for resection (e.g. tumor), cortical mapping (including awake) or intracranial electrode implantation
* Step 2: patients with pharmaco-resistant epilepsy hospitalized in the epilepsy monitoring unit (EMU) for the purpose of intracranial EEG monitoring

Exclusion Criteria:

* Patients with increased risk of infection
* Pregnant or breast-feeding women
* Severe neuropsychiatric disorders
* Severe cognitive problems: the patients need to be able to understand instructions and provide consent
* Chronic headache disorders, such as migraine and related disorders, as well as trigeminal neuralgia
* Medical conditions contraindicating cranial surgery (e.g. skin disorders causing poor wound healing, blood or cardiac disorder requiring chronic anti-coagulation, osteomyelitis, active systemic infection, haemorrhagic disease, diabetes, hepatitis, any documented allergy to implantation material)
* Other chronic, unstable medical conditions that could interfere with subject participation
* Existing scalp lesions or skin breakdown
* Scalp infections
* Implanted neurosurgical devices that are incompatible with Epios leads, which may include DBS leads
* Subjects who are allergic to the anaesthetics used in the implantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-11-02 (Actual)

PRIMARY OUTCOMES:
Feasibility of inserting Epios Leads in step 1 | Through the length of Step 1, up to 24 weeks
  The primary outcome of step 1 is to assess the feasibility of inserting two different EEG electrode leads (tubular and flat) under the human scalp via the tunneling tools.
  Measurement parameter:
  Length of each incision measured in centimeters.
Feasibility of inserting Epios Leads in step 2 | Through the length of Step 2 , up to 1 year
  The primary outcome of step 2 is to assess the feasibility of inserting Leads tridents (either tubular or flat depending on the outcome from step 1) under the human scalp via the tunneling tools.
  Measurement parameter:
  Length of each incision measured in millimeters.
Safety assessed as number of adverse events related to study device compared to the total number of adverse events for Step 1 | Through the length of Step 1, up to 24 weeks
  Patients' safety monitoring is ensured along the clinical study in a descriptive manner. Safety criteria resulting or not in early device explantation have been established to monitor patients' safety.
Safety assessed as number of adverse events related to study device compared to the total number of adverse events for Step 2 | Through the length of Step 2 , up to 1 year
  Patients' safety monitoring is ensured along the clinical study in a descriptive manner. Safety criteria resulting or not in early device explantation have been established to monitor patients' safety.

SECONDARY OUTCOMES:
Capability of tubular leads to record subscalp EEG signals in Step 1 | Through the length of Step 1, up to 24 weeks
  The investigator will compare the absolute amplitude and derive a power spectrum to identify the power distribution in each recording.
Capability of flat leads to record subscalp EEG signals in Step 1 | Through the length of Step 1, up to 24 weeks
  The investigator will compare the absolute amplitude and derive a power spectrum to identify the power distribution in each recording.
Capability of Epios leads to record epileptiform EEG signals from the sub-scalp space in Step 2 | Through the length of Step 2 , up to 1 year
  The investigator will compare power spectra in different electrodes from sub-scalp and intracranial EEG.
  Measurement parameter:
  Signal-to-Noise Ratio (SNR) analysis for the subcutaneous electrodes leads compared to intracranial electrodes.

OTHER OUTCOMES:
Qualitative surgical feedback on the handling of the two EEG lead designs in Step 1 | Immediately after each single implantation and final assessment after 24 weeks
  Measurement Parameters:
  Questionnaires:
  * Insertion tunneling toolkit (tear-away sheaths and stylets) used (yes/no choice)
  * Number of tear-away sheaths used (open field)
  * Number of stylets used (open field)
Qualitative comparison of EEG recordings between the two leads designs in Step 1 | Immediately after each single implantation and final assessment after 24 weeks
  Measurement Parameter:
  Questionnaires
Qualitative comparison to parallel scalp and intracranial EEG in Step 2 | Up to 21 days
  Measurement parameter:
  Questionnaires
Quantitative comparison to parallel scalp and intracranial EEG in Step 2 | Up to 21 days
  Comparison of power spectra in different electrodes from subscalp and intracranial EEG.
  Measurement parameter:
  Signal-to-Noise Ratio (SNR) analysis for the subcutaneous electrodes leads compared to intracranial electrodes.
Calculation of number of false negatives in expert detection of seizures in sub-scalp EEG in Step 2 | Through the length of Step 2 , up to 1 year
Collection of clinical pain assessment in Step 2 | Through the length of Step 2 , up to 1 year
  Descriptive pain perception on a scale from 0 ( no pain) to 10 (pain max). Numeric rating scales (NRS) is used.

CONTACTS AND LOCATIONS:
Overall Officials: Maxime Baud, MD, PhD, Principal Investigator — Universitätklinik für Neurologie, Inselspital, Bern University Hospital
Locations (1):
- Universitätklinik für Neurologie, Inselspital, Bern University, Bern, Switzerland

REFERENCES:
- [Derived] van Maren E, Alnes SL, Ramos da Cruz J, Sobolewski A, Friedrichs-Maeder C, Wohler K, Barlatey SL, Feruglio S, Fuchs M, Vlachos I, Zimmermann J, Bertolote T, Z'Graggen WJ, Tzovara A, Donoghue J, Kouvas G, Schindler K, Pollo C, Baud MO. Feasibility, Safety, and Performance of Full-Head Subscalp EEG Using Minimally Invasive Electrode Implantation. Neurology. 2024 Jun 25;102(12):e209428. doi: 10.1212/WNL.0000000000209428. Epub 2024 Jun 6. PMID 38843489